CLINICAL TRIAL: NCT00094016
Title: Safety and Efficacy Evaluation of Two Doses of HFA-Propelled Beclomethasone Dipropionate (QVAR) Versus Placebo by Breath Operated and Metered Dose Inhalers in Mild to Moderate Asthmatic Children
Brief Title: Evaluation of Two Doses of QVAR by Breath Operated and Metered Dose Inhalers in Asthmatic Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IXR-302-25-197
Record Dates: First submitted 2004-10-08; First posted 2004-10-11 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

INTERVENTIONS:
Drug: beclomethasone dipropionate

SUMMARY:
The primary objective of this study is to compare the QVAR-Easi-Breathe 100 mcg/day and QVAR-Easi-Breathe 200 mcg/day with placebo relative to changes in forced expiratory volume in 1 second (FEV1) results following 12 weeks of treatment. Secondary objectives such as daily asthma symptoms scores (per week), morning peak expiratory flow (PEF) values, nocturnal awakening and utilization of rescue medication per day also will be evaluated. In addition, an exploratory evaluation will assess the comparability of the two devices (i.e., QVAR-Easi-Breathe versus QVAR-MDI) at the same dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children aged 5 through 11 years at the screening visit
* Documented clinical evidence of asthma (FEV1 = 65-90%)
* Ability to perform acceptable and reproducible spirometry per ATS guidelines
* Ability to perform PEF determinations
* Reversible bronchoconstriction as verified by >12% increase in FEV1
* Otherwise healthy children with clinically-acceptable medical history, physical examination, vital signs and clinical laboratory parameters within the acceptable ranges for asthma patients
* The parent or guardian must be willing to give written informed consent as well as the patient assent and be able to adhere to the dose and visit schedule.

Exclusion Criteria:

* Patients who have used inhaled corticosteroids within 30 days prior to the screening visit.
* Allergy or sensitivity to beclomethasone dipropionate (BDP) or to other components of the formulations used in the CTM
* Patients demonstrating an increase or decrease in FEV1 >20% between the screening and baseline visit.
* Patients who are unable to use a metered dose inhaler (MDI) without a spacer device.
* Patients requiring the use of >12 puffs per day of albuterol for any 3 consecutive days between the screening and baseline visits.
* Patients with evidence of growth retardation
* Patients who have been treated with methotrexate, cyclosporin, gold or other cytotoxic agents for the control of asthma or for a concurrent condition within the last 3 months.
* Patients who are receiving escalating doses of immunotherapy, oral immunotherapy or short course (rush) immunotherapy for rhinitis.
* Patients with evidence (on physical exam) of oropharyngeal candidiasis.
* Exposure to investigational drugs within 30 days prior to the screening visit
* Require continuous treatment with beta blockers MAO inhibitors, tricyclic antidepressants, anticholinergics, inhaled nedocromil or cromolyn, or nebulized therapy (excluding sponsor provided albuterol MDI)
* Inability to tolerate or unwillingness to comply with required washout periods for all applicable medications
* Treatment at any time for life-threatening asthmatic episodes (e.g., episodes requiring intubation and/or associated with the development of hypercapnia, hypoxia and seizures, etc.)
* Patients that have received any of the following treatments or met any of the following conditions within six weeks prior to the screening visit:

  * Oral or injectable corticosteroids
  * an upper respiratory tract infection and/or sinusitis associated with exacerbation of asthmatic symptoms
  * emergency room treatment or hospitalization for asthmatic symptoms.
* History and/or presence of any non-asthmatic acute or chronic lung disease, including but not limited to bronchitis (within the previous 6 months), emphysema, active tuberculosis, bronchiectasis or cystic fibrosis.
* Presence of any clinically-significant cardiovascular disease (including cardiac arrhythmias and uncontrolled hypertension), clinically-significant hepatic, renal, or endocrine dysfunction, stroke, uncontrolled diabetes, hyperthyroidism, convulsive disorders, neoplastic disease other than basal cell carcinoma, and significant psychiatric disease.
* History of glaucoma or cataracts
* Presence of systemic fungal, bacterial, viral or parasitic infections and/or ocular herpes simplex
* Unlikely to be compliant, take study medication as directed, complete the diary cards, or attend scheduled clinic visits as required.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440
Dates: Start 2004-10-31 (Actual); Primary Completion 2006-06-30 (Actual); Study Completion 2006-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (37):
  - Allergy and Asthma Specialists, Huntington Beach, California
  - Pediatric Care Medical Group, Huntington Beach, California
  - West Coast Clinical Trials, Long Beach, California
  - Southern California Research, Mission Viejo, California
  - Clinical Trials of Orange County, Inc., Orange, California
  - California Allergy & Asthma, Palmdale, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Integrated Research Group, Riverside, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy and Asthma Medical Group, Walnut Creek, California
  - Allergy & Asthma Care of Florida, Ocala, Florida
  - New Horizon's Health Research, Atlanta, Georgia
  - AeroAllergy Research Labs of Savanna, Inc, Savannah, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Family Allergy & Asthma Research Institute, Louisville, Kentucky
  - Perez-Betancourt Medical Clinic, Metairie, Louisiana
  - NorthEast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Research Institute, Plymouth, Minnesota
  - The Asthma and Allergy Center, Papillion, Nebraska
  - Asthma and Allergy Associates, PC, Ithaca, New York
  - St.Elizabeth's Children's Health Center, Utica, New York
  - Regional Allergy and Asthma Consultants, Asheville, North Carolina
  - Allergy & Respiratory Center, Canton, Ohio
  - Dayton Clinical Research Center, Dayton, Ohio
  - Dr. Santiago Reyes, Oklahoma City, Oklahoma
  - Allergy and Asthma Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy and Asthma Research Groups, Eugene, Oregon
  - Allergy, Asthma & Dermatology Research Center, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - The Allergy Asthma and Sinus Center, Knoxville, Tennessee
  - Pediatric Allergy/Immunology Assoc., Dallas, Texas
  - Pharmaceutical Research and Consulting, Inc., Dallas, Texas
  - Allergy and Asthma Associates, Houston, Texas
  - Virginia Adult & Pediatric Allergy & Asthma, Richmond, Virginia
  - Spokane Allergy and Asthma Clinical Research, Spokane, Washington
- Puerto Rico (2):
  - Centro Neumologia Pediatrica, Hato Rey
  - Ponce School of Medicine, Ponce